CLINICAL TRIAL: NCT05728463
Title: Single Incision Laparoscopic Cholecystectomy Compared with Conventional Laparoscopic Cholecystectomy, a Randomized Controlled Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-0533
Record Dates: First submitted 2023-02-05; First posted 2023-02-15 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-02

CONDITIONS: Cholecystectomy, Laparoscopic
Keywords: Single-incision laparoscopic cholecystectomy; Conventional laparoscopic cholecystectomy
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-incision laparoscopic cholecystectomy (Experimental): SILC was defined as laparoscopic surgery done through a single trans-umbilical incision
  Interventions: Procedure: Laparoscopic cholecystectomy
- Conventional laparoscopic cholecystectomy (Active Comparator): CLC was defined as three or four port surgery carried out with either French or American position.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy is defined as total or subtotal desection of the gallbladder laparoscopically.

SUMMARY:
Laparoscopic cholecystectomy has been accepted and is nowadays considered as the gold standard treatment of gallstones disease. Conventional laparoscopic cholecystectomy (CLC) was defined as three or four port surgery carried out with either French or American position. It reduced post-operative pain and shorten post-operative length of stay compared with open cholecystectomy in a great extent. Single-incision laparoscopic cholecystectomy (SILC) as a revolutionized surgery, the main reason for its widespread use being the following: less post-operative pain, faster recovery, better cosmetics and quicker return to full activities, all resulting in the improvement of post-operative quality of life. SILC uses the umbilicus as a natural orifice allowing easy access to peritoneal cavity, easy conversion to standard laparoscopy and its easy closure, has been widely introduced into the clinical practice for benign gallbladder diseases. SILC can easily hide the surgical scar inside the umbilicus, thus has better cosmetic effect. But the real clinical benefits for patients still remain a matter of debate. In the last 5 years, many studies on SILC have been published, trying to answer the question whether such a new approach is worthwhile or not and whether is safe and cost-effective.Based on the above controversy, we conduct a RCT comparing clinical and peri-operative outcomes, such as quality of life (QOL), of SILC and CLC with the intent to assess the actual indications of the single-incision approach.

ELIGIBILITY:
Inclusion Criteria:

* Benign gallbladder disease

Exclusion Criteria:

* Combined with liver cirrhosis (Child grade B and above)
* Upper abdominal surgical history;
* Gallbladder gangrene perforation;
* Changes in surgical plan (conversion to laparotomy,cholangiography, bile duct exploration, bile duct injury repair, abscess clearance, multivisceral resection.)
* patients and their families do not agree with the treatment lost follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Quality of life (time to return to normal life) | 2 years
  The quality of life of patients after operation was investigated by a unified SF-36 questionnaire.

SECONDARY OUTCOMES:
Cosmetic result | 2 years
  Evaluation of postoperative incisional scarring using the Vancouver Scar Scale.The scar was observed after pressing with a special glass sheet for 2 seconds. The highest score was 15 points, and the lowest score was 0 points. The higher the score, the more serious the scar situation.
Grade II or above incidence of complications | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daren Liu, MD, PhD, Study Director — Chief Physician
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No